CLINICAL TRIAL: NCT05942898
Title: When the Alarm Goes Off, You're Already Awake!
Brief Title: When the Alarm Goes Off, You're Already Awake
Status: Completed | Type: Observational
Sponsor: International Institute of Behavioral Medicines (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-02
Record Dates: First submitted 2023-07-02; First posted 2023-07-12 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Anxiety
Keywords: Behavioral Medicine; Anticipatory anxiety; Alarm; Work; Experiencing self; Remembering self
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The present study does not contain any intervention — The present study does not contain any intervention

SUMMARY:
This is a behavioral observational study aimed at evaluating the impact that anxiety exerts on working people at the moment of awakening in the morning. It consists of a short self-administered questionnaire which will be given to workers to complete. Relationships between workers' answers and anxiety will be evaluated.

DETAILED DESCRIPTION:
This is a behavioral observational study aimed at evaluating the impact that anxiety exerts on working people at the moment of awakening in the morning. Literature found out that anticipatory anxiety plays a key role as for awakening quality (experiencing self). This evaluation could change at the end of the working day due to biased memory effects (remembering self).

In Literature there are not studies which investigate the relationships between time to awakening before the alarm sounds and anxiety.

The study consists of a short self-administered questionnaire which will be given to workers to complete. In more details, the survey is made of five questions collecting information on type of work, people who use an alarm, time of awakening before the alarm goes off, feelings on the moment of awakening, and feelings as for the working day spent. Further, participants will have to complete an anxiety self-administered questionnaire on anxiety, and namely the Zung Self-Rating Anxiety Scale.

Descriptive statistics will be presented by taking into account the characteristics of the sample being investigated. Statistical correlations between workers' answers and anxiety will be also evaluated.

This study's usefulness relies on detecting on advance mood disorders (like anxiety is) and maladaptive behaviors, in order to build persons' positive routines (i.e. well-being) and improve their productive quality at work.

ELIGIBILITY:
Inclusion Criteria:

* Being workers (any type)
* Adult age
* Ability to understand the Italian language

Exclusion Criteria:

* People who do not use the alarm clock to wake up in the morning
* Refuse to adhere to the study

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Workers (any kind)
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Zung | At the specific time of the scale assessment
  Zung Self-Rating Anxiety Scale; score 20-80 with higher estimates indicating higher levels of anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Barbara Rocca, Calosso, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dunstan DA, Scott N. Norms for Zung's Self-rating Anxiety Scale. BMC Psychiatry. 2020 Feb 28;20(1):90. doi: 10.1186/s12888-019-2427-6. PMID 32111187